CLINICAL TRIAL: NCT03582995
Title: Root Coverage With Acellular Dermal Matrix and Bovine Derived Osseous Xenograft Using Either a Coronally Positioned Tunnel or Coronally Positioned Flap
Brief Title: Root Coverage With Acellular Dermal Matrix and Bovine Derived Osseous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Program Director, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.0467
Record Dates: First submitted 2018-06-13; First posted 2018-07-11 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flap Surgery for root coverage with Alloderm and xenograft (Active Comparator): Root coverage surgery using a flap technique
  Interventions: Procedure: Flap Surgery for root coverage with Alloderm and xenograft
- Tunnel Surgery for root coverage with Alloderm and xenograft (Experimental): Root coverage surgery using a tunnel technique
  Interventions: Procedure: Tunnel Surgery for root coverage with Alloderm and xenograft

INTERVENTIONS:
Procedure: Flap Surgery for root coverage with Alloderm and xenograft — A coronally positioned FLAP technique with AlloDerm® GBR and osseous xenograft will be used for root coverage
  Arms: Flap Surgery for root coverage with Alloderm and xenograft
Procedure: Tunnel Surgery for root coverage with Alloderm and xenograft — A coronally positioned TUNNEL technique with AlloDerm® GBR and osseous xenograft will be used for root coverage.
  Arms: Tunnel Surgery for root coverage with Alloderm and xenograft

SUMMARY:
The study will consist of a randomized controlled clinical study trial comparing the results of coronally positioned flap with AlloDerm GBR plus bovine derived xenograft versus coronally positioned tunnel with AlloDerm GBR plus bovine derived xenograft in approximately 30 patients (15 per group). All materials used in the study are FDA approved.

DETAILED DESCRIPTION:
Patients will be assigned to one of two treatment groups. In the positive control group, BX will be placed over the root and bone surface of the defect, covered with ADM GBR® and sutured using a continuous sling suture technique (line angle to line angle) with a Maxon 5-0, 3/8 circle 13 mm needle (Dodge et. al, 1998). The coronally positioned flap will be sutured separately and coronally positioned using a continuous sling suture technique (papilla to papilla sutures) with a Maxon 5-0, 3/8 circle 13 mm needle. In the test group, BX will be placed over the root and bone surface of the defect, covered with ADM GBR® and sutured together using a continuous sling suture technique (line angle to line angle) with a Maxon 5-0, 3/8 circle 13 mm needle. The coronally positioned tunnel will be sutured together and coronally positioned using a continuous sling suture technique (line angle to line angle) with a Maxon 5-0, 3/8 circle 13 mm needle.

Post-operative instructions will be given to the patients along with prescriptions, in appropriate cases, for systemic doxycycline 100 mg once a day for 14 days; an anti-inflammatory agent (naproxen 375 mg q12h for 7 days); an analgesic (hydrocodone/acetaminophen 5/325mg q6-8h prn pain); a steroid, Medrol dose pack, 21 tablets of 4 mg methylprednisolone; 6 tablets on day 1, 5 on day 2, decrease by 1/day until last tablet dose on day 6, or dexamethazone 1mg, 18 tablets, 3 tablets/day for 1st3 days, 2/day for the next 3 days, 1/day for the last 3 days (always taken in the morning).

All patients will be seen at week 1 or 2, 4, 8, 16 and 24, at which time the final exam will be completed. Sutures will be removed between weeks 4-8, as indicated. Post-operative visits will consist of supragingival plaque removal and oral hygiene reinforcement. Any patient who develops any adverse reaction to the materials used or shows attachment loss ≥2.0 mm will be exited from the study and will receive the appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

A. At least one Miller Class I or II mucogingival defect ≥ 3 mm (Miller 1985).

B. The mucogingival defect must be on a non-molar tooth.

C. Patients must be ≥ 18 years of age.

Exclusion Criteria:

A. Patients with debilitating systemic or diseases that significantly affect the periodontium.

B. Patients with a known allergy to any of the materials that will be used in the study, including systemic antibiotics (tetracycline and doxycycline).

C. Patients requiring antibiotic prophylaxis.

D. Root surface restorations at the site of recession.

E. No detectable CEJ

F. Patients who fail to maintain oral hygiene levels of at least 80% plaque free surfaces.

G. Patients who are pregnant or lactating.

H. Patients who use tobacco products (smoking or smokeless tobacco).

I. Patients with alcohol abuse problems.

J. Patients undergoing long-term steroid therapy.

K. History of previous root coverage procedures, graft or GTR, on the test teeth.

L. Patients who fail to complete the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage | 4 months
  Initial and final recession will be measured from the cementoenamel junction to the gingival margin in millimeters. Root coverage will be determined by the amount of initial recession minus the final recession. Percent root coverage will be determined by root coverage divided by initial recession, multiplied by 100

SECONDARY OUTCOMES:
Tissue thickness | 4 months
  The thickness of the gingival tissue will be

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MS, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics, UofL School of Dentistry, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No